CLINICAL TRIAL: NCT00476242
Title: Placebo Controlled Study of Memantine as an Adjunct to Naltrexone in the Treatment of Opioid Dependence
Brief Title: Memantine as a Supplement to Naltrexone in Treating Heroin Dependence
Acronym: NAMHS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5936R R01 DA015822-01; R01DA015822 (NIH); NCT00126711 (obsolete NCT alias)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Opioid Dependence; Heroin Dependence
Keywords: heroin abuse; opiate abuse; opioid dependence; naltrexone; memantine
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — vivitrol; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine and Vivitrol (Experimental): intramuscular injection of Vivitrol 380 mg and 20 mg bid Memantine (PO)
  Interventions: Drug: Vivitrol; Drug: memantine
- Placebo and Vivitrol (Placebo Comparator): intramuscular injection of Vivitrol 380 mg and Placebo
  Interventions: Drug: Vivitrol

INTERVENTIONS:
Drug: Vivitrol — intramuscular injection of Vivitrol 380 mg for up to 6 months (six injections)
  Other Names: intramuscular injection of Vivitrol 380 mg
Drug: memantine — Memantine will be given in two divided doses, starting with the second day of the naltrexone induction, with the target doses of 40 mg/day (or the maximum tolerated dose), for a total of twelve weeks of medication treatment.
  Arms: Memantine and Vivitrol

SUMMARY:
Prospective participants will undergo a screening process at the clinic to determine eligibility. After screening, eligible patients will complete an 8-day inpatient detoxification, followed by a 12-week outpatient phase. Patients will be randomly assigned to one of two conditions (1) Naltrexone + Placebo; (2) Naltrexone + Memantine 20 mg bid. Long-acting, injectable form of naltrexone (Vivitrol) will be administered once per month (the total of three injections) while memantine or placebo will be taken daily. In addition, patients will receive twice weekly psychosocial intervention that will include motivational interviewing and cognitive-behavioral relapse prevention. The outpatient treatment will also consist of 3 weekly visits to the clinic in which patients will receive counseling to help maintain abstinence and improve compliance with study medication.

DETAILED DESCRIPTION:
In the proposed trial heroin-dependent patients undergoing detoxification will be randomly assigned to one of two conditions (1) Naltrexone + Placebo; (2) Naltrexone + Memantine 20 mg bid. Long-acting, injectable form of naltrexone (Vivitrol) will be administered once per month (the total of three injections) while memantine or placebo will be taken daily. In addition, patients will receive twice weekly psychosocial intervention that will include motivational interviewing and cognitive-behavioral relapse prevention. The goal of psychosocial intervention is to improve compliance with medication and maintain abstinence. A double-blind trial will last twelve weeks with assessments at baseline and at each appointment three times per week. After the completion of a double-blind study (experimental phase), participants will continue open label treatment with Vivitrol and therapy for additional three months (study extension phase). Repeated assessments will also be completed one, two, and three months following the end of double-blind treatment. For the experimental phase of the study, the primary aim is to test the efficacy of memantine in reducing early attrition and improving outcome in opioid-dependent individuals maintained on naltrexone and primary outcome measures will be retention in treatment by the end of the study and heroin abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, aged 18-60.
2. Meets Diagnostic and Statistical Manual IV (DSM-IV) criteria for current opiate dependence disorder of at least six months duration, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear.
3. Able to give informed consent.

Exclusion Criteria:

1. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.
2. Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with serum glutamic oxaloacetic transaminase or serum glutamic-pyruvic transaminase levels >2 times normal, unstable diabetes, chronic organic mental disorder (e.g., AIDS dementia).
3. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV schizophrenia, bipolar disorder with mania or psychosis, and depressive disorder with suicide risk or 1 or more suicide attempts within the past year.
4. History of allergic reaction to buprenorphine, naloxone, memantine, naltrexone, clonidine, or clonazepam.
5. Currently prescribed or regularly taking opiates for chronic pain or medical illness.
6. Current participation in another intensive psychotherapy or substance abuse treatment program or currently prescribed psychotropic medications.
7. Current participation in a methadone maintenance treatment program and/or regular use of illicit methadone (>30 mg per week).
8. History of accidental drug overdose in the last three years or any other significant history of overdose following detoxification defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

REFERENCES:
- [Result] Bisaga A, Sullivan MA, Cheng WY, Carpenter KM, Mariani JJ, Levin FR, Raby WN, Nunes EV. A placebo controlled trial of memantine as an adjunct to oral naltrexone for opioid dependence. Drug Alcohol Depend. 2011 Dec 1;119(1-2):e23-9. doi: 10.1016/j.drugalcdep.2011.05.019. Epub 2011 Jun 28. PMID 21715107
- See also: stars website — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants dropped during the inpatient detoxification, therefore only 55 participants were randomized out of the 82 total enrolled.
Groups:
- Placebo and Vivitrol: Participants treated with placebo capsules and Vivitrol.
- Memantine and Vivitrol: Participants treated with memantine 40 mg/d capsules and Vivitrol.
Period: Overall Study
Arm/Group | Placebo and Vivitrol | Memantine and Vivitrol
Started | 27 | 28
Completed | 19 | 12
Not Completed | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine and Vivitrol | Placebo and Vivitrol | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (12.0) | 39.0 (11.5) | 39.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 24 | 20 | 44
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Opiate Use Measured by Urine Toxicology Results
Description: Opiate use was qualified by the number of opiate positive urine results.
Time Frame: 3x/week during 12 weeks of the trial or study participation
Measure: Median (Inter-Quartile Range); unit: Percent of total urine samples
Arm/Group | Memantine and Vivitrol | Placebo and Vivitrol
Number analyzed (Participants) | 28 | 27
Percent of total urine samples | 9 [3 to 40] | 10 [0 to 19]

2. Primary Outcome: Retention in Treatment The Primary Outcome Measure Will be the Dichotomous Measure Retention in Treatment (Whether the Patient Completes the 12 Week Trial, Yes/no).
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Memantine and Vivitrol | Placebo and Vivitrol
Number analyzed (Participants) | 28 | 27
participants | 12 | 19
Statistical Analysis 1: Comparison: Memantine and Vivitrol vs Placebo and Vivitrol; Test type: Superiority or Other; p = .047, Log Rank

3. Secondary Outcome: Opiate Craving Based on Heroin Craving Scale
Description: Range 0- 100 ( 0= no craving; 100= very strong craving
Time Frame: Average of twice weekly assessments for 12 weeks of study or length of participation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo and Vivitrol | Memantine and Vivitrol
Number analyzed (Participants) | 27 | 28
units on a scale | 18.47 (25.79) | 15.74 (22.22)

ADVERSE EVENTS:
Arm/Group | Memantine and Vivitrol | Placebo and Vivitrol
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27
Other Adverse Events (participants affected / at risk) | 20/28 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine and Vivitrol (N=28) | Placebo and Vivitrol (N=27)
Psychiatric worsening (Psychiatric disorders) | 1 | 0 — The participant attended two outpatient visits, and was removed from the study due to psychiatric worsening (irritability, insomnia, and disorganized thinking).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine and Vivitrol (N=28) | Placebo and Vivitrol (N=27)
Insomnia (Psychiatric disorders) | 17 (17) | 13 (13)
Mood changes (Psychiatric disorders) | 7 (7) | 9 (9)
Increased/decreased appetite (Psychiatric disorders) | 6 (6) | 5 (5)
Fatigue/drowsiness (Psychiatric disorders) | 7 (7) | 8 (8)
Nausea/Vomiting (Psychiatric disorders) | 1 (1) | 4 (4)
Diarrhea (Psychiatric disorders) | 7 (7) | 3 (3)
Headache (Psychiatric disorders) | 2 (2) | 4 (4)
Body Aches (Psychiatric disorders) | 4 (4) | 6 (6)
GI Distress (Psychiatric disorders) | 4 (4) | 7 (7)
Sweating/chills (Psychiatric disorders) | 2 (2) | 5 (5)
Faintness/dizziness (Psychiatric disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No